CLINICAL TRIAL: NCT05535725
Title: Single Blinded Randomized Clinical Trial on the Application of Powdered Vancomycin in the Surgical Wound as Prophylaxis Against the Occurrence of Surgical Site Infection at La Paix State University Hospital Haiti
Brief Title: Application of Powdered Vancomycin in the Surgical Wound in Haiti
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinique Ortos (Other)
Responsible Party: Principal Investigator, Augustin Delange Hendrick, principal investigator, Clinique Ortos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CliniqueOrtos 0590
Record Dates: First submitted 2022-08-07; First posted 2022-09-10 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Surgical Site Infection
Keywords: surgical site infection; vancomycin
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: the randomization sequence was created using Stata 9.0 ware statistical software and was stratified by center with a 1:1 allocation using random block sizes of 2, 4 and 6." "Participants were randomly assigned following simple randomization procedures to 1 of 2 treatment groups
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- expose (Experimental): A group of patients receiving 1g of powdered vancomycin in the operative wound before its closure, and another group not receiving it
  Interventions: Drug: application of powdered vancomycin in the surgical wound as prophylaxis against the occurrence of surgical site infection
- non expose (No Intervention): A group of patients not receiving 1g of powdered vancomycin in the operative wound before its closure

INTERVENTIONS:
Drug: application of powdered vancomycin in the surgical wound as prophylaxis against the occurrence of surgical site infection — on the application of powdered vancomycin in the surgical wound as prophylaxis against the occurrence of surgical site infection at La Paix State University Hospital Haiti over 2 years.Both groups benefited from the same preoperative asepsis protocol. One hour before the incision, 1g of intravenous ceftriaxone is administered to the patients, this dose is maintained during the 48 hours postoperative every 12 hours. At discharged the two groups of patients received oral cloxacilin 500mg three times a day for one week. Patients are dressed every 2 days until the surgical wound has healed. Patients are seen in the outpatient clinic at 2, 4, and 6 weeks, then at one year. We selected 215 patients and retained 204.
  Arms: expose

SUMMARY:
Vancomycin, a tricyclic glycopeptide antibiotic, was originally indicated for the treatment of penicillin-resistant S. Aureus. It has a bactericidal action, inhibiting the biosynthesis of the cell wall of Gram-positive bacteria. Various studies have reported the application of intraoperative vancomycin powder to the wound prior to wound closure as a method of antibiotic prophylaxis. Intrasite administration of the drug should theoretically minimize rapid absorption into the systemic circulation, thereby reducing drug-associated side effects. The precipitated concentration gradient between the local wound and the scaffold should also reduce the occurrence of drug resistance. In Haiti, monitoring patients post-operatively is often difficult. The Mortality, Morbidity and Use of Services Survey (EMMUS-VI 2016-2017) reports that the non-use of a health facility is motivated in 58% of cases by the excessively high economic cost of care. Also, SSIs represent a challenge for clinicians. The best solution to the consequences of SSI in this context is prevention. In the present study, the investigator tested the hypothesis that the use of vancomycin powder in the surgical wound would decrease the occurrence of SSI.

DETAILED DESCRIPTION:
Type of study

This is a single-center prospective study with balanced blind randomization 1: 1 in parallel group.

Method and materials

After approval of the research protocol by the hospital ethics committee, the randomization sequence will be created using Stata 9.0 ware statistical software and will be stratified by center with a 1:1 allocation using random block sizes of 2, 4 and 6." "Participants will be randomly assigned following simple randomization procedures to 1 of 2 treatment groups. A group of patients will receive 2g of powdered vancomycin in the operative wound before its closure, and another group will not receive it. Both groups will benefit from the same preoperative asepsis protocol. One hour before the incision, 1g of intravenous ceftriaxone will be administered to the patients, this dose is maintained during the 48 hours postoperative every 12 hours. At discharged the two groups of patients will receive oral cloxacilin 500mg three times a day for one week. Patients are dressed every 2 days until the surgical wound has healed. Patients will be seen in the outpatient clinic at 2, 4, and 6 weeks, then at one year.

The significance level for the statistical tests is 0.05%. investigator used chi-square tests to assess the degree of relationship. The frequency of the patient's demographic, clinical and therapeutic characteristics are calculated. We used pubmed, google scholar, medline to perform the literature review. The consort guide will be used for the methodology.

ELIGIBILITY:
Inclusion Criteria:

* patients with 18 years and older
* lower extremity fractures

Exclusion Criteria:

* patients with impaired consciousness,
* those with an open Gustillo and Anderson type III fracture
* those with a C reactive protein > 6.
* those with date of trauma more than 48 hours
* those with passage of purulent secretion in the wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Crossover between ISOs and the two study groups | 12 month
  Crossover Chi Square between ISOs and the two study groups. the significant value of p=0.005.
age | 12 month
  age: quantitative variable the age written on the national identification card Average age =(sum of study ages)/(number of study patients)
sexe | 12 month
  this variable is qualitative and has three modalities 1) male 2) female 3) orther frequency sex X = Number of cases of X / number of total cases Sexeratio=(majority sex)/(minority sex)
origin | 12 month
  qualitative variable. the place where the patient lives. frequency origin X = Number of cases of X / number of total cases this variable has 2 modalities: 1 patient from the capital 2) patient from outside of the capital
comorbidity | 12 month
  qualitative variable. Association of two diseases, mental or physical, frequently observed in the population frequency comorbidity X = Number of cases of X / number of total cases
habits | 12 month
  qualitative variable. mores, customs, customs specific to the patient frequency comorbidity X = Number of cases of X / number of total cases this variable has 2 modalities 1) alcoholic 2)smoker
type of surgery | 12 month
  the surgical technique used this variable qualitative has 6 modality (nail, plate, prothesis, DHS, pinning, vissage, cerclage) frequency X = Number of cases of X / number of total cases
Timing of the surgery | 12 month
  the surgical timing :the time elapsed between the incision and the closure of the skin this variable qualitative has 3 modality ; Less than 1 h ;1 to 2h ; More than 2h
  frequency X = Number of cases of X / number of total cases

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Orthos, Port-au-Prince, Haiti

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calderone RR, Garland DE, Capen DA, Oster H. Cost of medical care for postoperative spinal infections. Orthop Clin North Am. 1996 Jan;27(1):171-82. PMID 8539047
- [Background] Graf K, Ott E, Vonberg RP, Kuehn C, Schilling T, Haverich A, Chaberny IF. Surgical site infections--economic consequences for the health care system. Langenbecks Arch Surg. 2011 Apr;396(4):453-9. doi: 10.1007/s00423-011-0772-0. Epub 2011 Mar 15. PMID 21404004
- [Background] Sweet FA, Roh M, Sliva C. Intrawound application of vancomycin for prophylaxis in instrumented thoracolumbar fusions: efficacy, drug levels, and patient outcomes. Spine (Phila Pa 1976). 2011 Nov 15;36(24):2084-8. doi: 10.1097/BRS.0b013e3181ff2cb1. PMID 21304438
- [Background] Zebala LP, Chuntarapas T, Kelly MP, Talcott M, Greco S, Riew KD. Intrawound vancomycin powder eradicates surgical wound contamination: an in vivo rabbit study. J Bone Joint Surg Am. 2014 Jan 1;96(1):46-51. doi: 10.2106/JBJS.L.01257. PMID 24382724
- [Background] O'Neill KR, Smith JG, Abtahi AM, Archer KR, Spengler DM, McGirt MJ, Devin CJ. Reduced surgical site infections in patients undergoing posterior spinal stabilization of traumatic injuries using vancomycin powder. Spine J. 2011 Jul;11(7):641-6. doi: 10.1016/j.spinee.2011.04.025. Epub 2011 May 19. PMID 21600853
- [Background] Molinari RW, Khera OA, Molinari WJ 3rd. Prophylactic intraoperative powdered vancomycin and postoperative deep spinal wound infection: 1,512 consecutive surgical cases over a 6-year period. Eur Spine J. 2012 Jun;21 Suppl 4(Suppl 4):S476-82. doi: 10.1007/s00586-011-2104-z. Epub 2011 Dec 8. PMID 22160172